CLINICAL TRIAL: NCT01326416
Title: Evaluation of the Impact of Physical Reconditioning Associated With Specific Nutritional Supplementation in Obese Patients Suffering From Metabolic Syndrome. OBEFITT Study.
Brief Title: Evaluation of the Impact of Physical Reconditioning Associated With Specific Nutritional Supplementation in Obese Patients Suffering From Metabolic Syndrome
Acronym: OBEFITT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/066/HP
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: obesity; metabolic syndrome; leucine; arginine; physical activity
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Motor Activity | interventions — Leucine; Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- S: Nutritional Supplementation alone (Active Comparator): Specific nutritional supplementation for six months by 30g per day of a mixture of amino acids (21 g of L-Leucine and 9 g of L-arginine), to distribute during each of the 3 main meals.
  Interventions: Dietary Supplement: L-Leucine and L-arginine
- A: Physical Reconditioning alone (Active Comparator): Physical reconditioning sessions led by a trainer three times a week for 6 months.
  Interventions: Other: Physical Reconditioning by a trainer
- AS: Physical Reconditioning + Nutritional Supplementation (Active Comparator): Association for six months of a specific nutritional supplementation by 21 g of L-Leucine and 9 g of L-arginine per day (to distribute during each of the 3 main meals) and of physical reconditioning sessions three times a week.
  Interventions: Other: Physical Reconditioning by a trainer
- C: Lifestyle counseling (No Intervention): Usual advice given in consultation on the need for a balanced diet and regular physical activity

INTERVENTIONS:
Dietary Supplement: L-Leucine and L-arginine — Specific nutritional supplementation for six months by 30g per day of a mixture of amino acids (21 g L-Leucine and 9 g of L-arginine), to be distributed during each of the 3 main meals.
  Arms: S: Nutritional Supplementation alone
Other: Physical Reconditioning by a trainer — Physical reconditioning sessions begin with a warm-up for five minutes for the type of effort made, and then correspond to a sporting course composed of elements of strength training and / or aerobic exercises and will be completed by a return to simple stretching and general advice on managing their physical life. The duration of each session will be 45 minutes at the beginning of the protocol and then gradually increased over time to achieve 1:30 of total physical activity at the end of protocol.
  Arms: A: Physical Reconditioning alone; AS: Physical Reconditioning + Nutritional Supplementation

SUMMARY:
Android obesity contributes, via insulin resistance and endothelial dysfunction, to the development of cardiovascular atherosclerosis. It leads to poor quality of life. It is often associated with metabolic syndrome which includes, whatever the definitions used (National Education Cholesterol Program, NECP / Adult Treatment Panel III, ATP III or International Diabetes Federation, IDF), an increased waist measurement, an arterial high blood pressure and disorders of the glucide and lipid metabolism. The treatment of the current "epidemic" of obesity and metabolic syndrome in France (12.4 % of obese and 14 % of subjects with metabolic syndrome) thus requires new therapeutic approaches.

A well-balanced diet and a daily physical activity are the indispensable requirements for the treatment of obesity and metabolic syndrome. It is possible to associate it to pharmacological agents, but the results are often partial and transient. Preliminary data suggest that leucine or arginine supplementation could facilitate the loss of fat mass. Moreover, the physical exercise has also demonstrated benefits.

Sessions of physical reconditioning (aerobic work + muscular intensification) associated with a program of specific nutritional supplementation by a mixture of Leucine and Arginine (in the daytime) could improve the treatment of obese subjects affected by metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from obesity (Body Mass Index (BMI) > 30kg.m-2) with a maximal weight of 135 kg
* Suffering from metabolic syndrome (International Federation of Diabetes(FID) definition)
* Hospitalized or followed in consultation
* Age 18 to 55 years old
* Not having recently participated in other clinical studies during the last days before pre-inclusion consultation
* Affiliated to a National Insurance scheme
* Having National Social Security insurance

Exclusion Criteria:

* Asthma, chronic respiratory failure, obstructive chronic bronchitis
* Current or recent Pneumothorax, recent pleural draining or biopsy, current hemoptysis, untreated / in course of treatment active tuberculosis
* Coronaropathy, myocardiopathy, myocarditis, unstable cardiac failure, ventricular rhythm disorders
* Severe Anemia
* Severe inferior members Arteritis
* Incapacity to walk or cycle
* Severe renal failure (Creatinine Clearance <or = 30 mL/min)
* Severe Sepsis
* Psychiatric Disorders (Diagnostic and Statistical Manual - Revision 4 (DSM IV) criteria) such as schizophrenia, other psychoses or major depressive non treated syndromes
* Severe or non treated Eating Disorders implicated in obesity (compulsive access, bulimia)
* Patients under guardianship or with curators
* Women in age of procreation without means of effective contraception
* Pregnant or breast-feeding women
* Taking medicates such as: proteinate powder (Protifar ®, SP95 ®, Orlistat (Xenical ®, Ally ®), exenatide (Byetta ®), sitagliptin (Januvia ®, Xelevia ®), vildagliptin (Galvus ®), sitagliptin-metformin (Janumet ®), Vildagliptin-metformin (Eucreas ®), tadalafil (Cialis ®) sildenafil (Viagra ®)
* Drug addiction to opiates in the last six months
* Alcohol or drug abuse
* Infection by Human Immunodeficiency Virus (HIV) , viral hepatitis B and viral hepatitis C
* Active addiction to smoking in more than 8 cigarettes a day
* Understanding badly spoken or written French
* Performed, in 2 to 3 days preceding the Dual-energy X-Ray Absorptiometry (DEXA) exam, of a bone scintigraphy or a digestive tract radiological examination with the use of barium type of contrast agent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2011-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Total body fat mass | 6 months
  Change in total body fat mass estimated by Dual-energy X-Ray Absorptiometry (DEXA).

SECONDARY OUTCOMES:
Weight | 6 months
  Change in weight, visceral fat mass, total lean mass, Bone Mineral Density, clinical and biological parameters of metabolic syndrome, insulin resistance, vascular inflammation parameters, heart rate variability, quadriceps strength, ventilatory parameters and quality of life score.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa FOLOPE, M.D., Principal Investigator — University Hospital, Rouen
Locations (1):
- University Hospital of Rouen, Rouen, France